CLINICAL TRIAL: NCT06107413
Title: A Phase 2, Randomized Study to Evaluate Safety, Efficacy, and Optimal Dose of ABBV-400 in Combination With Fluorouracil, Folinic Acid, and Bevacizumab and to Evaluate Safety and Efficacy of ABBV-400 in Combination With Bevacizumab in Previously Treated Subjects With Unresectable Metastatic Colorectal Cancer
Brief Title: Study to Assess Adverse Events and Change in Disease Activity in Previously Treated Adult Participants Receiving Intravenous (IV) ABBV-400 With Unresectable Metastatic Colorectal Cancer in Combination With IV Fluorouracil, Folinic Acid, and Bevacizumab
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M24-311; 2023-505110-14 (Other: EU CT)
Record Dates: First submitted 2023-10-25; First posted 2023-10-30 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Unresectable Metastatic Colorectal Cancer
Keywords: Unresectable Metastatic Colorectal Cancer; ABBV-400; Fluorouracil; Folinic Acid; Bevacizumab; Cancer
MeSH Terms: conditions — Neoplasms | interventions — Bevacizumab; Leucovorin; Fluorouracil; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- Stage 1: ABBV-400+FFB A (Experimental): Participants will receive escalating ABBV-400 in combination with Fluorouracil, Folinic Acid, and Bevacizumab (FFB) on dose schedule A as part of the safety lead in, during the 3 year study duration.
  Interventions: Drug: ABBV-400; Drug: Bevacizumab; Drug: Folinic Acid; Drug: Fluorouracil
- Stage 1: ABBV-400+FFB B (Experimental): Participants will receive escalating ABBV-400 in combination with FFB on dose schedule B as part of the safety lead in, during the 3 year study duration.
  Interventions: Drug: ABBV-400; Drug: Bevacizumab; Drug: Folinic Acid; Drug: Fluorouracil
- Stage 2: ABBV-400+FFB A Low (Experimental): Participants will receive ABBV-400 in combination with FFB at the low dose determined in the safety lead in on dose schedule A as part of the dose optimization, during the 3 year study duration.
  Interventions: Drug: ABBV-400; Drug: Bevacizumab; Drug: Folinic Acid; Drug: Fluorouracil
- Stage 2: ABBV-400+FFB A High (Experimental): Participants will receive ABBV-400 in combination with FFB at the high dose determined in the safety lead in on dose schedule A as part of the dose optimization, during the 3 year study duration.
  Interventions: Drug: ABBV-400; Drug: Bevacizumab; Drug: Folinic Acid; Drug: Fluorouracil
- Stage 2: FFB+Irinotecan (Standard of Care [SOC]) (Experimental): Participants will receive SOC during the 3 year study duration.
  Interventions: Drug: Bevacizumab; Drug: Folinic Acid; Drug: Fluorouracil; Drug: Irinotecan
- Stage 3: ABBV-400+FFB B Low (Experimental): Participants will receive ABBV-400 in combination with FFB at the low dose determined in the safety lead in on dose schedule A as part of the dose optimization/expansion, during the 3 year study duration.
  Interventions: Drug: ABBV-400; Drug: Bevacizumab; Drug: Folinic Acid; Drug: Fluorouracil
- Stage 3: ABBV-400+Bevacizumab C High (Experimental): Participants will receive ABBV-400 in combination with Bevacizumab at the high dose determined in the safety lead in on dose schedule C as part of the dose optimization/expansion, during the 3 year study duration.
  Interventions: Drug: ABBV-400; Drug: Bevacizumab

INTERVENTIONS:
Drug: ABBV-400 — Intravenous (IV) Infusion
  Arms: Stage 1: ABBV-400+FFB A; Stage 1: ABBV-400+FFB B; Stage 2: ABBV-400+FFB A High; Stage 2: ABBV-400+FFB A Low; Stage 3: ABBV-400+Bevacizumab C High; Stage 3: ABBV-400+FFB B Low
Drug: Bevacizumab — IV Infusion
Drug: Folinic Acid — IV Infusion
  Arms: Stage 1: ABBV-400+FFB A; Stage 1: ABBV-400+FFB B; Stage 2: ABBV-400+FFB A High; Stage 2: ABBV-400+FFB A Low; Stage 2: FFB+Irinotecan (Standard of Care [SOC]); Stage 3: ABBV-400+FFB B Low
Drug: Fluorouracil — IV Infusion
  Arms: Stage 1: ABBV-400+FFB A; Stage 1: ABBV-400+FFB B; Stage 2: ABBV-400+FFB A High; Stage 2: ABBV-400+FFB A Low; Stage 2: FFB+Irinotecan (Standard of Care [SOC]); Stage 3: ABBV-400+FFB B Low
Drug: Irinotecan — IV Infusion
  Arms: Stage 2: FFB+Irinotecan (Standard of Care [SOC])

SUMMARY:
Cancer is a condition where cells in a specific part of body grow and reproduce uncontrollably. The purpose of this study is to assess adverse events and change in disease activity when ABBV-400 is given in combination with Fluorouracil, Folinic Acid, and Bevacizumab to adult participants to treat unresctable metastatic colorectal cancer.

ABBV-400 is an investigational drug being developed for the treatment of unresectable metastatic colorectal cancer. Fluorouracil, folinic acid, and bevacizumab (FFB) is an approved drug for the treatment of unresectable metastatic colorectal cancer. Study doctors put the participants in groups called treatment arms. Each treatment arm receives a different dose of ABBV-400 in combination with FFB in escalating doses on two different schedules (safety lead in), followed by low or high doses of ABBV-400 in combination with FFB or fluorouracil, folinic acid, irinotecan, and bevacizumab (standard of care [SOC]) [dose optimization] on its own, ending with low or high doses of ABBV-400 in combination with FFB for continued dose optimization and expansion. Approximately 280 adult participants with unresectable metastatic colorectal cancer will be enrolled in the study in 65 sites worldwide.

In the safety lead in, participants will receive escalating intravenous (IV) ABBV-400 in combination with IV FFB on two different schedules. During the dose optimization participants will receive IV ABBV-400 in combination with IV FFB at low or high doses determined in the safety lead in. The dose optimization arm will also include a comparator cohort in which participants will receive SOC. During the dose optimization and expansion stage, participants will receive IV ABBV-400 in combination with IV FFB at low or high doses that have been determined from the previous stages. The study will run for a duration of approximately 3 years.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at an approved institution (hospital or clinic). The effect of the treatment will be frequently checked by medical assessments, blood tests, questionnaires and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histologically or cytologically confirmed unresectable metastatic colorectal cancer (mCRC).
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
* Progressed on only one first-line (1L) systemic treatment of combination chemotherapy in the metastatic setting with or without targeted therapy.

Exclusion Criteria:

* Harbor the BRAF V600E mutation.
* dMMR+/MSI-H.
* Received anticancer therapy including chemotherapy, radiation therapy, immunotherapy, biologic, or any investigational therapy within 28 days or 5 half-lives of the drug (whichever is shorter) prior to the first dose of ABBV-400.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2023-11-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Objective Response | Up to 24 Weeks
  OR is defined as complete response (CR) or partial response (PR) as assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1, as assessed by the investigator.
Progression Free Survival (PFS) | Up to 11 Months
  PFS is defined as the time from the first dose of study drug to the first occurrence of radiographic progression based on RECIST version 1.1 as determined by the investigator or death from any cause, whichever occurs earlier.
Number of Participants with Adverse Events (AEs) | Up to 3 Years
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Duration of Response (DOR) | Up to 7 Months
  DOR is defined as The time from the first documented CR or PR to the first occurrence of radiographic progression per RECIST v1.1 as determined by the investigator or death from any cause, whichever occurs first.
Overall Survival (OS) | Up to 3 Years
  OS is defined as the time from first dose of study drug to the event of death from any cause.
Percentage of Participants Achieving Best Overall Response (BOR) | Up to 18 Weeks
  BOR is defined as confirmed CR or confirmed PR, or stable disease (SD) based on RECIST, version 1.1 as determined by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (64):
- United States (22):
  - Mayo Clinic Arizona /ID# 262610, Phoenix, Arizona
  - Highlands Oncology Group, PA /ID# 259424, Springdale, Arkansas
  - City of Hope National Medical Center /ID# 257576, Duarte, California
  - City of Hope - Orange County Lennar Foundation Cancer Center /ID# 268365, Irvine, California
  - Yale School of Medicine /ID# 257494, New Haven, Connecticut
  - Mayo Clinic Hospital Jacksonville /ID# 262609, Jacksonville, Florida
  - University of Illinois Hospital and Health Sciences System /ID# 257300, Chicago, Illinois
  - Northwestern Medicine - Northwestern Memorial Hospital /ID# 260563, Chicago, Illinois
  - Fort Wayne Medical Oncology and Hematology- South Office /ID# 259601, Fort Wayne, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center /ID# 258789, Indianapolis, Indiana
  - Community Health Network, Inc. /ID# 257078, Indianapolis, Indiana
  - Comprehensive Cancer Centers of Nevada /ID# 257642, Henderson, Louisiana
  - Mayo Clinic - Rochester /ID# 257301, Rochester, Minnesota
  - Atrium Health Levine Cancer Institute /ID# 258840, Charlotte, North Carolina
  - Duke Cancer Institute /ID# 257236, Durham, North Carolina
  - Oregon Health & Science University, Knight Cancer Institute- /ID# 259190, Portland, Oregon
  - Medical University of South Carolina /ID# 258486, Charleston, South Carolina
  - Avera Cancer Institute /ID# 257949, Sioux Falls, South Dakota
  - MD Anderson Cancer Center /ID# 258713, Houston, Texas
  - Texas Oncology PA /ID# 257780, Houston, Texas
  - Inova Schar Cancer Institute - Fairfax - Innovation Park Drive /ID# 257448, Fairfax, Virginia
  - Virginia Cancer Specialists - Fairfax /ID# 257261, Fairfax, Virginia
- Belgium (7):
  - Imelda Ziekenhuis /ID# 257082, Bonheiden, Antwerpen
  - Universitair Ziekenhuis Antwerpen /ID# 257080, Edegem, Antwerpen
  - Cliniques Universitaires UCL Saint-Luc /ID# 257081, Brussels, Brussels Capital
  - UZ Gent /ID# 257083, Ghent, Oost-Vlaanderen
  - Universitair Ziekenhuis Leuven /ID# 257079, Leuven, Vlaams-Brabant
  - AZ-Delta /ID# 257084, Roeselare, West-Vlaanderen
  - Institut Jules Bordet /ID# 257625, Anderlecht
- Germany (6):
  - Universitatsklinikum Mannheim /ID# 257781, Mannheim, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen /ID# 258780, Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Ulm /ID# 257783, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Carl Gustav Carus Dresden /ID# 257787, Dresden, Saxony
  - Charite Universitaetsmedizin Berlin Campus Virchow-Klinikum /ID# 257785, Berlin
  - Universitaetsklinikum Hamburg-Eppendorf /ID# 257782, Hamburg
- Israel (7):
  - Meir Medical Center /ID# 257089, Kfar Saba, Central District
  - Shaare Zedek Medical Center /ID# 259253, Jerusalem, Jerusalem
  - Hadassah /ID# 257088, Jerusalem, Jerusalem
  - The Chaim Sheba Medical Center /ID# 257312, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 257090, Tel Aviv, Tel Aviv
  - Rambam Health Care Campus /ID# 257344, Haifa
  - Assuta Medical Center /ID# 267581, Tel Aviv
- Japan (5):
  - Aichi Cancer Center Hospital /ID# 257286, Nagoya, Aichi-ken
  - National Cancer Center Hospital East /ID# 257282, Kashiwa-shi, Chiba
  - Kyoto University Hospital /ID# 257287, Kyoto, Kyoto
  - Shizuoka Cancer Center /ID# 257288, Sunto-gun, Shizuoka
  - National Cancer Center Hospital /ID# 257284, Chuo-ku, Tokyo
- South Korea (5):
  - Chonnam National University Hwasun Hospital /ID# 258366, Hwasun-gun, Jeonranamdo
  - Seoul National University Hospital /ID# 257493, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 257845, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 257571, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 257492, Seoul
- Spain (6):
  - Hospital Universitario Vall de Hebron /ID# 257383, Barcelona
  - Hospital General Universitario Gregorio Maranon /ID# 257387, Madrid
  - Hospital Universitario 12 de Octubre /ID# 257384, Madrid
  - Hospital Universitario HM Sanchinarro /ID# 258549, Madrid
  - Hospital Clinico Universitario de Valencia /ID# 257385, Valencia
  - Hospital Universitario Miguel Servet /ID# 257388, Zaragoza
- Taiwan (6):
  - Kaohsiung Chang Gung Memorial Hospital /ID# 257675, Kaohsiung City, Kaohsiung
  - National Taiwan University Hospital /ID# 257639, Taipei City, Taipei
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 257637, Kaohsiung City
  - National Cheng Kung University Hospital /ID# 257638, Tainan
  - Taipei Veterans General Hosp /ID# 257636, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 257640, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-311